CLINICAL TRIAL: NCT05875376
Title: Establish the Couple Intervention Program for Adults With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202106091RINC
Record Dates: First submitted 2023-04-14; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder, couple therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASD couple (Experimental): Either one of the couple has ASD diagnosis, including couples who are married or in romantic relationship.
  Interventions: Behavioral: Couple group therapy

INTERVENTIONS:
Behavioral: Couple group therapy — 1. Introduction of "I" statements
  2. Focus of each conversation
  3. Emotion acknowledgement
  4. Self-assurance and positive feedback
  5. teamwork and cooperation
  6. Reflection

SUMMARY:
The development of adult intimate relationships and the transition into couplehood are part of most people's life cycles, but these transitions become very challenging for individuals diagnosed with autism spectrum disorder (ASD) in as much as social interactions, emotional communication, and reciprocity, which are essential for interpersonal relationships, are made more difficult due to the condition itself. In the Adult ASD Clinic of National Taiwan University Hospital, we observe that the wives of the ASD husband suffer from long-term frustration, loneliness and helplessness, and are frequently experience anxiety and depression, that in turns changes the family's function and impacts on children's mental health. To date, there are limited intervention models focusing on couple therapy for ASD adults (or neurodiverse couple). Given the strong needs of clinical service, this study aims to identify the common problems of the ASD couples and develop a program to improve their partner relationships.

ELIGIBILITY:
Inclusion Criteria:

* one person of each couple has either Autism Spectrum Disorder diagnosis or the autism spectrum quotient scoring above or equal to 26
* able to communicate in Chinese
* Wechsler Intelligence scoring above 70

Exclusion Criteria:

* Psychiatric disorder (i.e. schizophrenia, substance abuse)
* unable to communication (i.e. visual or auditory impairment)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Autism Diagnostic Observation Schedule, ADOS | 6 weeks
  range from 0 to 8 for each item. Higher the score, worse the symptoms
Autism Spectrum Quotient | 6 weeks
  range from 0 to 3 for each item, total score of 50. Higher the score, wrose the related symptoms.
Empathy Quotient | 6 weeks
  range from 0 to 3 for each item, total score of 40. Higher the score, worse the empathy
Social Responsiveness Scale, SRS | 6 weeks
  65 questions, range from 1 to 5. Higher the score, worse the symptom
Quality of socialization questionnaire, QSQ | 6 weeks
  selected part of the questionnaire to examine the quality of interaction. Higher the score, better the socialization

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan